CLINICAL TRIAL: NCT05689554
Title: Reducing CNS-Active Medications to Prevent Falls and Injuries in Older Adults
Acronym: STOP-FALLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Elizabeth Phelan, Professor, Division of Gerontology & Geriatric Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SITE00000971; CD002967 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC))
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aging; Accidental Fall

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Educational intervention
  Interventions: Behavioral: STOP Falls Educational Intervention
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: STOP Falls Educational Intervention — This is a pragmatic, cluster-randomized, parallel-group, controlled clinical trial. The unit of randomization is the clinic, to avoid the risk of contamination if healthcare providers within a clinic were randomized (i.e., reducing the potential for intervention providers to communicate with control providers about the intervention and share materials). Eighteen clinics were identified for the trial, of which 9 were randomized to the intervention and 9 to usual care.
  Arms: Intervention

SUMMARY:
The overall objective of STOP-FALLS is to test whether a patient-centered deprescribing intervention that focuses on CNS-active medications reduces medically treated falls among older adults. The aims are: AIM 1: Adapt and pilot-test an evidence-based medication reduction intervention for use in an integrated health care system. AIM 2: Implement and evaluate the adapted intervention using a cluster-randomized controlled trial design. Aim 3: Assess barriers and facilitators to intervention implementation.

DETAILED DESCRIPTION:
Background: Central nervous system (CNS) active medications have been consistently linked to falls in older people. However, few randomized trials have evaluated whether CNS-active medication reduction reduces falls and fall-related injuries. The objective of the Reducing CNS-active Medications to Prevent Falls and Injuries in Older Adults (STOP-FALLS) trial is to test the effectiveness of a health-system-embedded deprescribing intervention focused on CNS-active medications on the incidence of medically treated falls among community-dwelling older adults.

This is a pragmatic, cluster-randomized, parallel-group, controlled clinical trial within Kaiser Permanente Washington to test the effectiveness of a 12-month deprescribing intervention consisting of: 1) an educational brochure and self-care handouts mailed to older adults prescribed one or more CNS-active medications (aged 60+: opioids, benzodiazepines and Z-drugs; aged 65+: skeletal muscle relaxants, tricyclic antidepressants, and antihistamines) and 2) decision support for their primary health care providers. Outcomes are examined over 18-26 months post-intervention. The primary outcome is first incident (post-baseline) medically treated fall as determined from health plan data. Sample size calculations ensured at least 80% power to detect a 20% reduction in the rate of medically treated falls for participants receiving care within the intervention (n=9) versus usual care clinics (n=9) assuming 18 months of follow-up. Secondary outcomes include medication discontinuation or dose reduction of any target medications. Safety outcomes include serious adverse drug withdrawal events, unintentional overdose, and death. The study team will also examine medication signetur fields for attempts to decrease medications. The study team will report factors affecting implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* For opioid and sedative-hypnotic medications, eligible participants are aged 60 years or older, while for skeletal muscle relaxants, tricyclic antidepressants, and first-generation antihistamines, eligible participants are aged 65 years or older.

Eligible participants must be long-term users of the target medication, defined as pharmacy dispensing of at least one of the target medication classes for at least 70 of the prior 90 days.

Further, eligible participants must either be assigned to a primary care provider (PCP) or have had 1+ visits in the prior year with a PCP at one of the 18 Kaiser Permanente Washington clinics participating in the study.

Exclusion Criteria:

1. diagnosis of dementia or a prescription for a medication used to treat dementia (i.e., a cholinesterase inhibitor or memantine);
2. residence in a skilled nursing facility;
3. metastatic cancer diagnosis in the prior 12 months;
4. receiving hospice or palliative care;
5. legally blind (unable to read print materials);
6. indication the participant requires a translator (cannot read materials printed in English); g) enrolled in other KPWA opioid deprescribing research studies;

h) enrolled in a KPWA pharmacy-driven initiative to reduce opioid doses; or i) diagnosed with opioid use disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2367 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Phelan, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Phelan EA, Williamson BD, Balderson BH, Cook AJ, Piccorelli AV, Fujii MM, Nakata KG, Graham VF, Theis MK, Turner JP, Tannenbaum C, Gray SL. Reducing Central Nervous System-Active Medications to Prevent Falls and Injuries Among Older Adults: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2424234. doi: 10.1001/jamanetworkopen.2024.24234. PMID 39052289
- [Derived] Balderson BH, Gray SL, Fujii MM, Nakata KG, Williamson BD, Cook AJ, Wellman R, Theis MK, Lewis CC, Key D, Phelan EA. A health-system-embedded deprescribing intervention targeting patients and providers to prevent falls in older adults (STOP-FALLS trial): study protocol for a pragmatic cluster-randomized controlled trial. Trials. 2023 May 11;24(1):322. doi: 10.1186/s13063-023-07336-7. PMID 37170329

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinic
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 1106; 9 Clinic | 1261; 9 Clinic
Completed | 1106; 9 Clinic | 1261; 9 Clinic
Not Completed | 0; 0 Clinic | 0; 0 Clinic

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual care
  Those receiving usual care and no intervention
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 1106 | 1261 | 2367
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 245 | 282 | 527
  >=65 years | 861 | 979 | 1840
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.4) | 70.9 (7.7) | 70.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 704 | 784 | 1488
  Male | 402 | 477 | 879
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 40 | 78
  Not Hispanic or Latino | 1068 | 1221 | 2289
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 11 | 29
  Asian | 16 | 21 | 37
  Native Hawaiian or Other Pacific Islander | 8 | 4 | 12
  Black or African American | 38 | 30 | 68
  White | 957 | 1099 | 2056
  More than one race | 24 | 32 | 56
  Unknown or Not Reported | 45 | 64 | 109

OUTCOME MEASURES:

1. Primary Outcome: Medically Treated Falls
Description: Falls for which medical attention is sought
Time Frame: up to 26 months following intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 1106 | 1261
Participants | 328 | 349
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.11, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [.944 to 1.306]

2. Secondary Outcome: Medication Discontinuation
Description: Target medication has not been prescribed for 90 days 6 months post intervention
Time Frame: 6 months following intervention
Population: Number of participants who were not prescribed the target medication of interest 90 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 1106 | 1261
Participants
  Opioids | 32 | 40
  Benzodiazepines | 55 | 49
  Tricyclic Antidepressants | 34 | 23
  Muscle Relaxants | 34 | 40
  Antihistamines (rx) | 5 | 0
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.183, Regression, modified Poisson; Risk Ratio (RR) = 1.24, 95% CI 2-sided [.9 to 1.7]

ADVERSE EVENTS:
Time Frame: Events were collected 6 months after study enrollement
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 86/1106 | 72/1261
Serious Adverse Events (participants affected / at risk) | 10/1106 | 4/1261
Other Adverse Events (participants affected / at risk) | 0/1106 | 0/1261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=1106) | Usual Care (N=1261)
Serious adverse drug withdrawal events involving opioids or sedative-hypnotics (General disorders) | 10 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT05689554/Prot_SAP_001.pdf